CLINICAL TRIAL: NCT07002307
Title: The Effect of Honey-sweetened Coffee, Black Tea and Green Tea on Blood Pressure, Heart Rate and Blood Glucose
Brief Title: The Effect of Honey-sweetened Coffee, Black Tea and Green Tea on Some Physiological Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Uyo Teaching Hospital (Other)
Responsible Party: Principal Investigator, Esther Oluwasola Aluko, Principal Investigator (PI), University of Uyo Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Uuthuyo
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Blood Pressure; Heart Rate; Blood Glucose
Keywords: Coffee; Honey-sweetened coffee; Black tea; Honey-sweetened black tea; Green Tea; Honey-sweetened green tea; Blood pressure; Heart rate; Blood glucose
MeSH Terms: interventions — Coffee; Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Control group (Placebo Comparator): Will receive 250 mL of warm water
  Interventions: Other: Warm water at 35 oC
- Coffee group (Active Comparator): Will receive 2.25 g of coffee dissolved in 250 mL of hot water
  Interventions: Other: Coffee
- Honey-sweetened coffee group (Active Comparator): Will receive 2.25 g of coffee plus 20 mL of honey put in 250 mL of hot water
  Interventions: Other: Honey-sweetened coffee
- Green tea group (Active Comparator): Will receive 2 g of green tea infuse in 250 mL of hot water
  Interventions: Other: Green tea
- Honey-sweetened green tea group (Active Comparator): Will receive 2 g of green tea plus 250 mL of honey put in 250 mL of hot water
  Interventions: Other: Honey-sweetened green tea
- Black tea group (Active Comparator): Will receive 2 g of black tea infuse in 250 mL of hot water
  Interventions: Other: Black tea
- Honey-sweetened black tea group (Active Comparator): Will receive 2 g of black tea plus 20 mL of honey put in 250 mL of hot water
  Interventions: Other: Honey-sweetened black tea

INTERVENTIONS:
Other: Warm water at 35 oC — The placebo for the control group
  Arms: Control group
Other: Coffee — Instant coffee, Nescafé Gold Blend, manufactured by Nestlé Coffee Brand, Nestlé Global
  Arms: Coffee group
Other: Honey-sweetened coffee — Instant coffee plus raw dark amber honey produced by Apis mellifera adansonii
  Arms: Honey-sweetened coffee group
Other: Green tea — Qualitea Natural Green Tea, packed by Qualitea Ceylon (PVT) LTD
  Arms: Green tea group
Other: Honey-sweetened green tea — Green tea plus honey
  Arms: Honey-sweetened green tea group
Other: Black tea — Lipton Yellow Label Black Tea
  Arms: Black tea group
Other: Honey-sweetened black tea — Black tea plus honey
  Arms: Honey-sweetened black tea group

SUMMARY:
The goal of this clinical trial is to investigate whether a three-day consumption of honey-sweetened black tea, green tea, and coffee will have an effect on blood pressure, heart rate, and blood glucose. The main questions it aims to answer are:

Does honey-sweetened black tea, green tea, and coffee, respectively, have the ability to influence blood pressure, heart rate, or blood glucose level?

Research will compare honey-sweetened black tea, green tea, and coffee to a placebo (warm water) to see if honey-sweetened black tea, green tea, and coffee work to reduce or increase blood pressure, heart rate, or blood glucose.

Participants will:

Take honey-sweetened black tea, green tea, and coffee, OR plain black tea, green tea, and coffee, OR warm water, one cup a day for 3 days The beverages will be taken at the Physiology laboratory, University of Uyo, and the participants will be observed for 60 minutes, during which their blood pressure, heart rate, and blood glucose level will be measured. This procedure will be repeated for the 3 days of study.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria are as follows:

* Age between 18 and 26
* Non-habitual coffee and tea drinkers who consume coffee, green tea, or black tea 2-5 times in the last two months
* Non-allergic to coffee, green tea, black tea, or honey
* Absence of medication use
* Will refrain from ingesting energy drinks, carbonated beverages, caffeinated beverages, or food for 24 hours before the study and throughout the study periods
* Will not consume anything except water after 11 p.m. during the experimental days Will be available and cooperate throughout the study duration.

Exclusion Criteria:

Exclusion criteria are as follows:

* Presence of cardiovascular disorders, hypertension, or diabetes
* Blood pressure above 120/80 mmHg and random blood glucose above 125 mg/dL
* Alcohol intake
* Smoking
* Habitual coffee or tea drinker

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Will be measured before consumption of the beverages and at 15, 30, 45, and 60 minutes after consumption of the beverages. This procedure will be repeated for 3 consecutive days.
Heart rate | Will be measured before consumption of the beverages and at 15, 30, 45, and 60 minutes after consumption of the beverages. This procedure will be repeated for 3 consecutive days.
Blood glucose | Will be measured before consumption of the beverages and at 30 and 60 minutes after consumption of the beverages. This procedure will be repeated for 3 consecutive days.

SECONDARY OUTCOMES:
Age | Will obtained during the eligibility process
Height | Will be measured on the first day of the experiment before the commencement of the experiment.
Body weight | Measurements will be taken over the course of the 3-day study prior to the commencement of the experiment each day.

CONTACTS AND LOCATIONS:
Overall Officials: Esther O Aluko, Principal Investigator — University of Uyo
Locations (1):
- Physiology laboratory, Physiology Department, Faculty of Basic Medical Sciences, University of Uyo, Uyo, Akwa Ibom State, Nigeria

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-05-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT07002307/Prot_SAP_ICF_000.pdf